CLINICAL TRIAL: NCT00874614
Title: A Phase II Study Evaluating the Efficacy and Safety of Ultratrace Iobenguane I 131 in Patients With Malignant Relapsed/Refractory Pheochromocytoma/Paraganglioma
Brief Title: A Study Evaluating Ultratrace Iobenguane I131 in Patients With Malignant Relapsed/Refractory Pheochromocytoma/Paraganglioma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Molecular Insight Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIP-IB12B
Expanded Access: NCT02961491 (Approved for marketing)
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Results first posted 2018-10-05 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Pheochromocytoma; Paraganglioma
Keywords: radiotherapy; MIBG; Azedra; neuroendocrine tumors; Iobenguane I 131; progenics
MeSH Terms: conditions — Pheochromocytoma; Paraganglioma; Neuroendocrine Tumors | interventions — 3-Iodobenzylguanidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ultratrace® Iobenguane I 131 Treatment (Experimental)
  Interventions: Radiation: Ultratrace® Iobenguane I131

INTERVENTIONS:
Radiation: Ultratrace® Iobenguane I131 — Each subject will be administered 3 mCi to 6 mCi Ultratrace® Iobenguane I 131, referred to as the Imaging Dose, to confirm that subject meets radiological entry criteria and to establish dosimetry. All subjects meeting entry criteria will then receive the investigational product referred to as the Therapeutic Dose (500 mCi or 8 mCi/kg if the subject weighs 62.5 kg or less) of Ultratrace Iobenguane I 131, followed by imaging at 7 days post infusion or upon discharge from isolation. The Therapeutic Doses will be adjusted equally if warranted by results of the dosimetry evaluation. At least 3 months later, subjects will receive the second Therapeutic Dose.
  Other Names: Azedra®; MIBG

SUMMARY:
This clinical trial is designed to evaluate the effectiveness and collect additional safety information on AZEDRA® (iobenguane I 131) for the treatment of metastatic or relapsed/refractory (to other treatment) or unresectable pheochromocytoma or paraganglioma.

The purpose of this trial is to test the use of AZEDRA® as a treatment for pheochromocytoma and paraganglioma, a rare disease. This Phase II study will help determine primarily if using the drug reduces the amount of blood pressure medication being taken as a result of the cancer and secondarily to determine such things as the effectiveness of the study drug in treating the cancer, additional safety measures, and to assess if the drug helps the quality of life and use of pain medication. All subjects will receive an imaging dose with scans followed by two therapeutic doses given approximately 3 months apart.

DETAILED DESCRIPTION:
AZEDRA® (Iobenguane I 131) is a very high-specific-activity iobenguane I 131, produced using proprietary Ultratrace® platform. Based on the well-characterized cellular active transport mechanism, the high specific activity of allows for effective cellular uptake of radioactivity and hence greater tumor uptake.

During this study the subjects will receive two (2) Therapy Doses that are given approximately three (3) months apart. Prior to administration of the first Therapy Dose, subjects will be given an Imaging Dose of AZEDRA® and will undergo iobenguane I 131 scans to evaluate tumor uptake and to measure normal organ distribution and allow for the calculation of radiation dose to normal organs.

Screening procedures for eligibility will need to be done before imaging or therapeutic doses of AZEDRA® are administered.

Hospitalization is required for approximately one (1) week after each of the two (2) Therapeutic Doses. Frequent follow up is necessary for the first year and some of the follow up visits may be done by a visiting health care professional in the subjects' homes. Subjects will be followed in the treatment study for one (1) year and for an additional four (4) years in long-term follow up.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 12 years of age
* Have a documented (medical record) diagnosis of either pheochromocytoma or paraganglioma
* Be ineligible for curative surgery for pheochromocytoma
* Have failed a prior therapy for pheochromocytoma/paraganglioma or are not candidates for chemotherapy or other curative therapies
* Be on stable antihypertensive medication for pheochromocytoma-related hypertension for at least 30 days
* Have at least one tumor site by CT or MR or iobenguane I 131 scan
* Have an expected survival of at least 6 months
* Subjects must agree to use an acceptable form of birth control (abstinence, IUD, oral contraception, barrier and spermicide or hormonal implant) during this study and for 6 months following Therapeutic Doses of Ultratrace Iobenguane I 131.
* Male subjects must agree not to father a child during the period beginning immediately after administration of the first Therapeutic Dose of Ultratrace Iobenguane I 131 during the study and ending six months after administration of the last Therapeutic Dose of Ultratrace Iobenguane I 131.

Exclusion Criteria:

Subjects will be excluded if any of the following conditions are observed:

* <50% of FDG (if data are available) positive lesions are MIBG avid
* Pregnant or nursing females
* Active CNS lesions by CT/MR scanning within 3 months of study entry
* New York Heart Association class IV heart failure, symptomatic congestive heart failure [New York Heart Association class IV with another medical disorder], unstable angina pectoris, cardiac arrhythmia
* Received any previous systemic radiotherapy resulting in marrow toxicity within 3 months of study entry or have active malignancy (other than pheochromocytoma/paraganglioma) requiring additional treatment during the active phase or follow up period of the Ultratrace® iobenguane I 131 trial.
* Administered prior whole-body radiation therapy
* Received external beam radiotherapy to > 25% of bone marrow
* Administered prior chemotherapy within 30 days or have active malignancy (other than pheochromocytoma/ paraganglioma) requiring additional treatment during the active phase or follow up period of the Ultratrace iobenguane I 131 trial.
* Karnofsky Performance Status is < 60
* Platelets < 80,000/μL
* Absolute neutrophil count (ANC) < 1,200/μL, Total bilirubin > 1.5 times the upper limit of normal, AST/SGOT or ALT/SGPT > 2.5 times the upper limit of normal
* Diagnosed with AIDS or HIV-positive
* Active chronic alcohol abuse, chronic liver disease or hepatitis
* Renal dysfunction/impairment
* Known allergy to iobenguane that has required medical intervention
* Received a therapeutic investigational compound and/or medical device/prior chemotherapy within 30 days before admission into this study
* Receiving a medication which inhibits tumor uptake of iobenguane I 131
* Any medical condition or other circumstances (i.e., uncontrolled current illness including but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with the study requirements.
* Any other condition, that in the opinion of the investigator, may compromise the safety or compliance of the subject or would preclude the subject from successful completion of the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2009-06-04 (Actual); Primary Completion 2017-02-14 (Actual); Study Completion 2021-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bennett Chin, MD, Principal Investigator — Duke University; Daniel Pryma, MD, Principal Investigator — University of Pennsylvania; Jeffrey Olsen, MD, Principal Investigator — Mallinckrodt Institute of Radiology Washington University; Camillo Jimenez, MD, Principal Investigator — MD Anderson Cancer; Joseph Dillon, MD, Principal Investigator — University of Iowa; Lilja Solnes, MD, Principal Investigator — Johns Hopkins University; Lale Kostakoglu, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Michael H Pampaloni, MD, Principal Investigator — University of California at San Francisco
Locations (10):
- United States (10):
  - University of California-San Francisco, San Francisco, California
  - University of Miami Miller School of Medicine, Miami, Florida
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins University, Baltimore, Maryland
  - Washington University School of Medicine, Alvin J. Siteman Cancer Center, St Louis, Missouri
  - Mount Sinai School of Medicine, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jimenez C, Chin BB, Noto RB, Dillon JS, Solnes L, Stambler N, DiPippo VA, Pryma DA. Biomarker response to high-specific-activity I-131 meta-iodobenzylguanidine in pheochromocytoma/paraganglioma. Endocr Relat Cancer. 2023 Jan 5;30(2):e220236. doi: 10.1530/ERC-22-0236. Print 2023 Feb 1. PMID 36472300

RESULTS

PARTICIPANT FLOW:
Groups:
- AZEDRA® (Iobenguane I 131): Patients received dosimetric dose (~5 mCi) of AZEDRA® via intravenous injection to confirm iobenguane-avidity and to establish dosimetry and biodistribution assessment. Eligible patients received a therapeutic dose of AZEDRA® based on body weight and reduced, if necessary, based on the dosimetry data. The second therapeutic dose is administered intravenously at least 90 days later.
Period: Overall Study
Arm/Group | AZEDRA® (Iobenguane I 131)
Started | 74
Received at Least One Therapeutic Dose | 68
Received Two Therapeutic Doses | 50
Completed (Completed or continuing in long-term follow-up phase) | 16 (As of December 2017)
Not Completed | 58

BASELINE CHARACTERISTICS:
Arm/Group | AZEDRA® (Iobenguane I 131)
Number analyzed (Participants) | 68
Age, Continuous [Median (Full Range); unit: years] | 55 [16 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 51
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Experienced a 50% or Greater Reduction (Including Discontinuation) of All Antihypertensive Medication(s) Lasting for at Least Six Months.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- AZEDRA® (Iobenguane I 131): Patients received at least one therapeutic dose of AZEDRA®.
Arm/Group | AZEDRA® (Iobenguane I 131)
Number analyzed (Participants) | 68
percentage of patients | 25 [16 to 37]

2. Secondary Outcome: Best Confirmed Overall Tumor Response of Complete Response (CR) or Partial Response (PR) by RECIST 1.0.
Description: Response Evaluation Criteria In Solid Tumors (RECIST) 1.0 was assessed by two independent central reviewers and one adjudicator, and overall response (PR or CR) was confirmed by follow-up imaging at the subsequent timepoint. Complete response was defined as confirmed disappearance of all target lesions and Partial Response was defined as confirmed decreased of >= 30% in baseline sum of the longest diameter of target lesions.
Time Frame: 12 months
Population: There were 64 patients with tumor measurements evaluable for tumor response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | AZEDRA® (Iobenguane I 131)
Number analyzed (Participants) | 64
percentage of patients | 23.4 [15 to 35]

3. Secondary Outcome: Changes From Baseline in Overall Quality of Life (QoL) - Best Response Within 12 Months After First Therapeutic Dose of AZEDRA®.
Description: The European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) C30 v.3 was used to evaluate QoL. This questionnaire was comprised of 30 questions, two of which pertain to a patient's Global Health Status and QoL. The two questions used a 7-point Likert scale of 1 (very poor) to 7 (excellent), in which the scores were averaged and linearly transformed to a 0-100 scale with higher scores indicating better health status and QoL. The questionnaire was administered at baseline and through 12 months after the first therapeutic dose of AZEDRA®. The results of QoL and changes from baseline were summarized by visit and the best response within 12 months after first therapeutic dose of AZEDRA® was reported. The outcome represents the mean change from baseline in overall QoL based on the best response reported within 12 months after first therapeutic dose of AZEDRA®.
Time Frame: 12 Months
Population: 53 patients with data available.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AZEDRA® (Iobenguane I 131)
Number analyzed (Participants) | 53
score on a scale | 17.5 (18.12)

4. Secondary Outcome: Overall Survival
Description: Duration of overall survival was calculated from the date of first therapeutic dose of AZEDRA® to death, or at the last date the patient was known to be alive. Results are presented per December 2017 data-cut. Survival was censored at the end of the 5-year long-term follow-up period, thus the upper limit of the confidence interval reported below for two therapeutic doses is actually >60 months.
Time Frame: Up to 5 Years (60 months)
Measure: Median (95% Confidence Interval); unit: months
Groups:
- At Least One Therapeutic Dose of AZEDRA®: Patients received at least one therapeutic dose of AZEDRA®.
- Two Therapeutic Doses of AZEDRA®: Patients received two therapeutic doses of AZEDRA®.
Arm/Group | At Least One Therapeutic Dose of AZEDRA® | Two Therapeutic Doses of AZEDRA®
Number analyzed (Participants) | 68 | 50
months | 37 [31 to 49] | 44 [32 to 60]

ADVERSE EVENTS:
Time Frame: All adverse events were collected from time of signed informed consent until the end of 15 weeks after the last therapeutic dose of AZEDRA®. Serious adverse events and adverse events of special interest were collected as part of long-term follow-up.
Groups:
- AZEDRA® (Iobenguane I 131): Patients who received any dose of AZEDRA® (N=74). All-cause mortality was followed in patients who received at least one therapeutic dose of AZEDRA® (N=68), up through long-term follow-up as of December 2017.
Arm/Group | AZEDRA® (Iobenguane I 131)
All-Cause Mortality (participants affected / at risk) | 31/68
Serious Adverse Events (participants affected / at risk) | 32/74
Other Adverse Events (participants affected / at risk) | 69/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZEDRA® (Iobenguane I 131) (N=74)
Thrombocytopenia (Blood and lymphatic system disorders) | 12
Anemia (Blood and lymphatic system disorders) | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Leukopenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 3
Sickle cell anemia with crisis (Blood and lymphatic system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Convulsion (Nervous system disorders) | 1
Dyskinesia (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Spinal cord compression (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Kidney fibrosis (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Cardiomyopathy (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Cellulitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Tendon injury (Injury, poisoning and procedural complications) | 1
Aspartate aminotransferase increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Mental status changes (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Hypertensive crisis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Disease progression (General disorders) | 1
Cholangitis acute (Hepatobiliary disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Spinal instability (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZEDRA® (Iobenguane I 131) (N=74)
Nausea (Gastrointestinal disorders) | 53
Vomiting (Gastrointestinal disorders) | 36
Dry mouth (Gastrointestinal disorders) | 28
Constipation (Gastrointestinal disorders) | 16
Diarrhea (Gastrointestinal disorders) | 16
Abdominal pain (Gastrointestinal disorders) | 14
Retching (Gastrointestinal disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 49
Anemia (Blood and lymphatic system disorders) | 43
Leukopenia (Blood and lymphatic system disorders) | 41
Neutropenia (Blood and lymphatic system disorders) | 39
Lymphopenia (Blood and lymphatic system disorders) | 10
Fatigue (General disorders) | 41
Asthenia (General disorders) | 14
Pyrexia (General disorders) | 9
Dizziness (Nervous system disorders) | 28
Headache (Nervous system disorders) | 21
Syncope (Nervous system disorders) | 4
White blood cell count decreased (Investigations) | 12
International normalized ratio increased (Investigations) | 11
Neutrophil count decreased (Investigations) | 10
Aspartate aminotransferase increased (Investigations) | 9
Hemoglobin decreased (Investigations) | 7
Platelet count decreased (Investigations) | 6
Alanine aminotransferase increased (Investigations) | 5
Hypotension (Vascular disorders) | 18
Hypertension (Vascular disorders) | 13
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4
Petechiae (Skin and subcutaneous tissue disorders) | 6
Decreased appetite (Metabolism and nutrition disorders) | 17
Dehydration (Metabolism and nutrition disorders) | 9
Tachycardia (Cardiac disorders) | 7
Contusion (Injury, poisoning and procedural complications) | 4
Salivary gland pain (Gastrointestinal disorders) | 10
Dyspepsia (Gastrointestinal disorders) | 8
Abdominal distension (Gastrointestinal disorders) | 5
Dysphagia (Gastrointestinal disorders) | 4
Edema peripheral (General disorders) | 9
Infusion site pain (General disorders) | 6
Injection site pain (General disorders) | 6
Chills (General disorders) | 5
Chest pain (General disorders) | 4
Dysgeusia (Nervous system disorders) | 13
Paraesthesia (Nervous system disorders) | 4
Weight decreased (Investigations) | 11
Prothrombin time prolonged (Investigations) | 8
Lymphocyte count decreased (Investigations) | 6
Blood alkaline phosphatase increased (Investigations) | 5
Blood creatinine increased (Investigations) | 5
Red blood cell count decreased (Investigations) | 5
Hematocrit decreased (Investigations) | 4
Sialoadenitis (Infections and infestations) | 14
Urinary tract infection (Infections and infestations) | 8
Candida infection (Infections and infestations) | 5
Upper respiratory tract infection (Infections and infestations) | 5
Nasopharyngitis (Infections and infestations) | 4
Sinusitis (Infections and infestations) | 4
Orthostatic hypotension (Vascular disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 11
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9
Neck pain (Musculoskeletal and connective tissue disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 8
Dry skin (Skin and subcutaneous tissue disorders) | 7
Alopecia (Skin and subcutaneous tissue disorders) | 4
Dermatitis contact (Skin and subcutaneous tissue disorders) | 4
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 4
Insomnia (Psychiatric disorders) | 7
Anxiety (Psychiatric disorders) | 4
Palpitations (Cardiac disorders) | 8
Proteinuria (Renal and urinary disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2014-03-21): https://cdn.clinicaltrials.gov/large-docs/14/NCT00874614/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-06): https://cdn.clinicaltrials.gov/large-docs/14/NCT00874614/SAP_001.pdf